CLINICAL TRIAL: NCT05530564
Title: Effect of Low-pressure Pneumoperitoneum on Pain and Inflammation in Laparoscopic Cholecystectomy: A Prospective Randomized Clinical Trial
Brief Title: Effect of Low-pressure Pneumoperitoneum on Pain and Inflammation in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Hanan Ibrahim Mansour, Dr. Hanan Mansour, M.D., University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10/2019/1115
Record Dates: First submitted 2022-08-27; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Pneumoperitoneum; Pain; Inflammatory Response
Keywords: Clinical trial; low pressure insufflation; pneumoperitoneum; laparoscopic cholecystectomy; pain; inflammatory marker
MeSH Terms: conditions — Pneumoperitoneum; Pain

STUDY DESIGN:
Intervention Model Description: participants were divided into two masked groups, labelled red and green; those operated at low-pressure pneumoperitoneum (green-label) and those operated at standard-pressure pneumoperitoneum (red-label).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: none of the participants knew at which pressure they will be operated on, nor the physicians who followed participants at floor or those analyzing blood samples, not the assigned physician to collect data, nor the personnel doing the analysis.
  only the operating surgeon and circulating nurse were aware of the meaning of the participant assigned label at time of operation. The masking was revealed post completion of analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-pressure pneumoperitoneum (Experimental): Participants undergone laparoscopic cholecystectomy by creation of a low-pressure pneumoperitoneum, set at 8-10 mm Hg
  Interventions: Procedure: low-pressure pneumoperitoneum
- Standard-pressure pneumoperitoneum (Active Comparator): Participants undergone laparoscopic cholecystectomy by creation of a standard-pressure pneumoperitoneum, set at 12-14 mm Hg
  Interventions: Procedure: standard-pressure pneumoperitoneum

INTERVENTIONS:
Procedure: low-pressure pneumoperitoneum — insufflation of the abdomen for creation of pneumoperitoneum, pressure set points between 8 to 10 mm Hg
  Arms: Low-pressure pneumoperitoneum
Procedure: standard-pressure pneumoperitoneum — insufflation of the abdomen for creation of pneumoperitoneum, pressure set points between 12 to 14 mm Hg
  Arms: Standard-pressure pneumoperitoneum

SUMMARY:
The purpose of this study is to assess the effect of low-pressure pneumoperitoneum on post operative pain and inflammation in patients undergoing elective laparoscopic cholecystectomy by comparing it to standard practice.

DETAILED DESCRIPTION:
After obtaining informed consent from eligible study participants. patients were randomized into one of two masked groups, labelled red and green. The red-label group was operated at standard-pressure pneumoperitoneum, while the green-label group was operated at low-pressure pneumoperitoneum. Baseline blood samples were obtained pre-operatively for ten inflammatory markers, patients' demographics and intra-operative details collected, then post-operative pain and change in inflammatory markers were followed.

ELIGIBILITY:
Inclusion Criteria:

- Elective admission for laparoscopic cholecystectomy

Exclusion Criteria:

* Current or previous diagnosis of acute cholecystitis confirmed by ultrasound
* previous GI surgeries, except bariatric and anti-reflux surgeries
* Currently on immunosuppressant agents
* Pregnancy
* Breastfeeding
* Currently diagnosed with drug addiction
* American Society of Anesthesiologists (ASA) score 3 and more

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
assessment of pain with SPS-11 at 6hr post-op | pre-op to 6 hours post op
  measure difference in pain on the 11-point short pain scale (SPS-11) at 6-hour post-op compared to baseline at pre-op, minimum score of 0 , maximun score of 10
  = pain at 6 hour post op - pain at pre-op
change in IL-6 | pre op to 24 hours post -op
  measure differance of inflammatory marker from baseline
  = baseline value- post op value (calculated in pg/mL) post-op collected at 24 hours from end of surgery

SECONDARY OUTCOMES:
assessment of difficulty of surgery | start to end of the study, 1 year
  to measure difference in surgery difficulty between the two groups using a scale of 1; easy, 2; moderate, 3; difficult.
  analysis done using Chi-square cross table on SPSS V 1.0.0.1406
assessment of difference in operation time | start to end of the study, 1 year
  to look for difference in operation time between the two groups, calculated in minutes.
  analysis done using Student's 2-tailed t-test on SPSS V 1.0.0.1406

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University Hospital, Amman, Jubaiha, Jordan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Reynolds W Jr. The first laparoscopic cholecystectomy. JSLS. 2001 Jan-Mar;5(1):89-94. PMID 11304004
- [Background] Soper NJ, Stockmann PT, Dunnegan DL, Ashley SW. Laparoscopic cholecystectomy. The new 'gold standard'? Arch Surg. 1992 Aug;127(8):917-21; discussion 921-3. doi: 10.1001/archsurg.1992.01420080051008. PMID 1386505
- [Background] Hypolito OH, Azevedo JL, de Lima Alvarenga Caldeira FM, de Azevedo OC, Miyahira SA, Miguel GP, Becker OM Jr, Machado AC, Nunes Filho GP, Azevedo GC. Creation of pneumoperitoneum: noninvasive monitoring of clinical effects of elevated intraperitoneal pressure for the insertion of the first trocar. Surg Endosc. 2010 Jul;24(7):1663-9. doi: 10.1007/s00464-009-0827-2. Epub 2009 Dec 25. PMID 20035347
- [Background] Ozdemir-van Brunschot DM, van Laarhoven KC, Scheffer GJ, Pouwels S, Wever KE, Warle MC. What is the evidence for the use of low-pressure pneumoperitoneum? A systematic review. Surg Endosc. 2016 May;30(5):2049-65. doi: 10.1007/s00464-015-4454-9. Epub 2015 Aug 15. PMID 26275545
- [Background] Gohil A. Comparison of low pressure versus standard pressure pneumoperitoneum for elective laparoscopic cholecystectomy in a tertiary care institute of western India. Int Surg J. 2018;5(5):1776. doi:10.18203/2349-2902.isj20181569
- [Background] Celarier S, Monziols S, Francois MO, Assenat V, Carles P, Capdepont M, Fleming C, Rullier E, Napolitano G, Denost Q. Randomized trial comparing low-pressure versus standard-pressure pneumoperitoneum in laparoscopic colectomy: PAROS trial. Trials. 2020 Feb 22;21(1):216. doi: 10.1186/s13063-020-4140-7. PMID 32087762
- [Background] Bhattacharjee HK, Jalaludeen A, Bansal V, Krishna A, Kumar S, Subramanium R, Ramachandran R, Misra M. Impact of standard-pressure and low-pressure pneumoperitoneum on shoulder pain following laparoscopic cholecystectomy: a randomised controlled trial. Surg Endosc. 2017 Mar;31(3):1287-1295. doi: 10.1007/s00464-016-5108-2. Epub 2016 Jul 21. PMID 27444831
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Background] Neudecker J, Sauerland S, Neugebauer E, Bergamaschi R, Bonjer HJ, Cuschieri A, Fuchs KH, Jacobi Ch, Jansen FW, Koivusalo AM, Lacy A, McMahon MJ, Millat B, Schwenk W. The European Association for Endoscopic Surgery clinical practice guideline on the pneumoperitoneum for laparoscopic surgery. Surg Endosc. 2002 Jul;16(7):1121-43. doi: 10.1007/s00464-001-9166-7. Epub 2001 May 20. PMID 12015619
- [Background] Hua J, Gong J, Yao L, Zhou B, Song Z. Low-pressure versus standard-pressure pneumoperitoneum for laparoscopic cholecystectomy: a systematic review and meta-analysis. Am J Surg. 2014 Jul;208(1):143-50. doi: 10.1016/j.amjsurg.2013.09.027. Epub 2014 Jan 16. PMID 24503370
- [Background] Mandal A, Ghosh A, Bakshi S. Low pressure versus standard pressure pneumoperitoneum in laparoscopic cholecystectomy: a comparative study. Int Surg J. 2020;7(5):1551. doi:10.18203/2349-2902.isj20201868
- [Background] Mahajan S, Shankar M, Garg VK, Gupta V, Sorout J. Intraoperative safety of low pressure pneumoperitoneum cholecystectomy: a comparative study. Int Surg J. 2017;4(11):3679. doi:10.18203/2349-2902.isj20174885
- [Background] Nasajiyan N, Javaherfourosh F, Ghomeishi A, Akhondzadeh R, Pazyar F, Hamoonpou N. Comparison of low and standard pressure gas injection at abdominal cavity on postoperative nausea and vomiting in laparoscopic cholecystectomy. Pak J Med Sci. 2014 Sep;30(5):1083-7. doi: 10.12669/pjms.305.5010. PMID 25225531
- [Background] Agarwal L, Kumawat S, Jain SA, Yadav A, Sharma S. Correlation of shoulder tip pain in case of low pressure and standard pressure pneumoperitoneum post laparoscopic cholecystectomy. Int Surg J. 2021;8(5):1522. doi:10.18203/2349-2902.isj20211820
- [Background] Barczynski M, Herman RM. A prospective randomized trial on comparison of low-pressure (LP) and standard-pressure (SP) pneumoperitoneum for laparoscopic cholecystectomy. Surg Endosc. 2003 Apr;17(4):533-8. doi: 10.1007/s00464-002-9121-2. Epub 2003 Feb 17. PMID 12582754
- [Background] Chang W, Yoo T, Cho WT, Cho G. Comparing postoperative pain in various pressure pneumoperitoneum of laparoscopic cholecystectomy: a double-blind randomized controlled study. Ann Surg Treat Res. 2021 May;100(5):276-281. doi: 10.4174/astr.2021.100.5.276. Epub 2021 Apr 29. PMID 34012945
- [Background] Moro ET, Pinto PCC, Neto AJMM, Hilkner AL, Salvador LFP, da Silva BRD, Souto IG, Boralli R, Bloomstone J. Quality of recovery in patients under low- or standard-pressure pneumoperitoneum. A randomised controlled trial. Acta Anaesthesiol Scand. 2021 Oct;65(9):1240-1247. doi: 10.1111/aas.13938. Epub 2021 Jun 24. PMID 34097759
- [Background] Dr. Vidyanand Tripathi, Dr. Angela B Marak, Dr. Resen Rajan S Methikkalam, Dr. Y Priyabarta Singh, Dr. S Tombisana, Prof. S Ranita Devi PGSM. A Comparative Study Between The Low Pressure Versus Standard Pressure Pneumoperitoneum In Laparoscopic Cholecyst... J Dent Med Sci. 2020;19(7):01-10. doi:10.9790/0853-1907140110
- [Background] Sodhi KS, Saxena AK, Ahuja CK, Rao K, Menon P, Kandelwal N. Postoperative appearances of esophageal atresia repair: retrospective study of 210 patients with review of literature - what the radiologist should know. Acta Radiol. 2013 Mar 1;54(2):221-5. doi: 10.1258/ar.2012.120274. Epub 2012 Nov 1. PMID 23117198
- [Background] Kanwer DB, Kaman L, Nedounsejiane M, Medhi B, Verma GR, Bala I. Comparative study of low pressure versus standard pressure pneumoperitoneum in laparoscopic cholecystectomy--a randomised controlled trial. Trop Gastroenterol. 2009 Jul-Sep;30(3):171-4. PMID 20306755
- [Background] Aggarwal M, Kumar A, Garg S, Pruthi A, Resident S. Effect of Low Pressure Versus High Pressure Pneumoperitoneum on Liver Functions in Laparoscopic Cholecystectomy. Int J Anat Radiol Surg. 2020;9(2):01-03
- [Background] Neogi P, Kumar P, Kumar S. Low-pressure Pneumoperitoneum in Laparoscopic Cholecystectomy: A Randomized Controlled Trial. Surg Laparosc Endosc Percutan Tech. 2020 Feb;30(1):30-34. doi: 10.1097/SLE.0000000000000719. PMID 31425453
- [Background] Schietroma M, Carlei F, Mownah A, Franchi L, Mazzotta C, Sozio A, Amicucci G. Changes in the blood coagulation, fibrinolysis, and cytokine profile during laparoscopic and open cholecystectomy. Surg Endosc. 2004 Jul;18(7):1090-6. doi: 10.1007/s00464-003-8819-0. Epub 2004 May 12. PMID 15136925
- [Background] Basgul E, Bahadir B, Celiker V, Karagoz AH, Hamaloglu E, Aypar U. Effects of low and high intra-abdominal pressure on immune response in laparoscopic cholecystectomy. Saudi Med J. 2004 Dec;25(12):1888-91. PMID 15711660
- [Background] Perrakis E, Vezakis A, Velimezis G, Savanis G, Deverakis S, Antoniades J, Sagkana E. Randomized comparison between different insufflation pressures for laparoscopic cholecystectomy. Surg Laparosc Endosc Percutan Tech. 2003 Aug;13(4):245-9. doi: 10.1097/00129689-200308000-00004. PMID 12960786
- [Background] Torres K, Torres A, Staskiewicz GJ, Chroscicki A, Los T, Maciejewski R. A comparative study of angiogenic and cytokine responses after laparoscopic cholecystectomy performed with standard- and low-pressure pneumoperitoneum. Surg Endosc. 2009 Sep;23(9):2117-23. doi: 10.1007/s00464-008-0234-0. Epub 2008 Dec 6. PMID 19067057
- [Background] Manou-Stathopoulou V, Korbonits M, Ackland GL. Redefining the perioperative stress response: a narrative review. Br J Anaesth. 2019 Nov;123(5):570-583. doi: 10.1016/j.bja.2019.08.011. Epub 2019 Sep 20. PMID 31547969
- [Background] Kwon YS, Jang JS, Hwang SM, Tark H, Kim JH, Lee JJ. Effects of surgery start time on postoperative cortisol, inflammatory cytokines, and postoperative hospital day in hip surgery: Randomized controlled trial. Medicine (Baltimore). 2019 Jun;98(24):e15820. doi: 10.1097/MD.0000000000015820. PMID 31192911
- [Background] Burton D, Nicholson G, Hall G. Endocrine and metabolic response to surgery. Contin Educ Anaesth Crit Care Pain. 2004;4(5):144-147. doi:10.1093/bjaceaccp/mkh040
- [Background] Chernow B, Alexander HR, Smallridge RC, Thompson WR, Cook D, Beardsley D, Fink MP, Lake CR, Fletcher JR. Hormonal responses to graded surgical stress. Arch Intern Med. 1987 Jul;147(7):1273-8. PMID 3606284
- [Background] Albers KI, Polat F, Panhuizen IF, Snoeck MMJ, Scheffer GJ, de Boer HD, Warle MC. The effect of low- versus normal-pressure pneumoperitoneum during laparoscopic colorectal surgery on the early quality of recovery with perioperative care according to the enhanced recovery principles (RECOVER): study protocol for a randomized controlled study. Trials. 2020 Jun 17;21(1):541. doi: 10.1186/s13063-020-04496-8. PMID 32552782
- [Background] Qin J, Song G, Jiang Y, Liu Q, Lin H. Low-pressure pneumoperitoneum reduces influence on ovarian hormones in infertile women: a randomised trial. Ann Palliat Med. 2021 May;10(5):5746-5753. doi: 10.21037/apm-21-476. Epub 2021 May 17. PMID 34044564
- [Background] Aditianingsih D, Mochtar CA, Lydia A, Siregar NC, Margyaningsih NI, Madjid AS, Suwarto S. Effects of low versus standard pressure pneumoperitoneum on renal syndecan-1 shedding and VEGF receptor-2 expression in living-donor nephrectomy: a randomized controlled study. BMC Anesthesiol. 2020 Feb 4;20(1):37. doi: 10.1186/s12871-020-0956-7. PMID 32019488
- [Derived] Rashdan M, Daradkeh S, Al-Ghazawi M, Abuhmeidan JH, Mahafthah A, Odeh G, Al-Qaisi M, Salameh I, Halaseh S, Al-Sabe L, Ahmad YB, Al-Ghazawi T, Al-Said M, Sha'bin S, Mansour H. Effect of low-pressure pneumoperitoneum on pain and inflammation in laparoscopic cholecystectomy: a randomized controlled clinical trial. BMC Res Notes. 2023 Sep 28;16(1):235. doi: 10.1186/s13104-023-06492-y. PMID 37770908

DOCUMENTS (2):
  • Study Protocol (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT05530564/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT05530564/SAP_001.pdf